CLINICAL TRIAL: NCT02036762
Title: EFFECTS OF RESPIRATORY MUSCLE STRETCH ON THORACOABDOMINAL MECHANIC, FUNCTIONAL CAPACITY, PSYCHOLOGICAL AND SOCIAL ASPECTS IN PATIENTS WITH CHRONIC OBSTRUCTIVE PULMONARY DISEASE
Brief Title: STRETCH OF RESPIRATORY MUSCLES IN PATIENTS WITH CHRONIC OBSTRUCTIVE PULMONARY DISEASE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Juliano Wada, Master Degree (in process), University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HCFMUSP 1295/09
Record Dates: First submitted 2013-08-15; First posted 2014-01-15 (Estimated); Last update posted 2014-01-15 (Estimated); Status verified 2014-01

CONDITIONS: Dyspnea; Quality of Life; Respiratory Symptoms
Keywords: Chronic Obstructive Pulmonary Disease; Thoracoabdominal Mechanics; Functional capacity; Quality of life
MeSH Terms: conditions — Dyspnea; Signs and Symptoms, Respiratory; Pulmonary Disease, Chronic Obstructive | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Group (Active Comparator): The group submitted to stretching exercises in the respiratory muscles and treadmill exercises
  Interventions: Other: Stretching Exercises
- Control Group (Sham Comparator): The control group received stretching exercises in the fist and ankle muscles and treadmill exercises
  Interventions: Other: Stretching Exercises

INTERVENTIONS:
Other: Stretching Exercises — The group submitted to stretching exercises in the respiratory muscles and treadmill exercises

SUMMARY:
THE AIM OF THIS STUDY IS TO TEST IF THE STRETCHING OF THE RESPIRATORY ACCESSORY MUSCLE PROVIDE SOME BENEFIT ON THORACOABDOMINAL MECHANICS, FUNCTIONAL CAPACITY, PSYCHOLOGICAL AND SOCIAL ASPECTS IN PATIENTS WITH CHRONIC OBSTRUCTIVE PULMONARY DISEASE

DETAILED DESCRIPTION:
PATIENTS WITH CHRONIC OBSTRUCTIVE PULMONARY DISEASE WILL BE SUBMITTED TO PASSIVE STRETCHING OF RESPIRATORY MUSCLES AND EXERCISE IN TREADMILL DURING 12 WEEKS, TWICE A WEEK. ONE WEEK AFTER THE TRAINING PERIOD, THE FUNCTIONAL CAPACITY, THE THORACOABDOMINAL MECHANICS AND LEVELS OF ANXIETY AND DEPRESSION WILL BE ASSESSED.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Obstructive Pulmonary Disease Diagnosis
* Clinical stability
* Absence of previous thoracic surgery
* Absence of other limitations

Exclusion Criteria:

* Copd exacerbation
* Absence greater than three days

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-11; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Functional Capacity | One week after the end of training
  Distance obtained (in meters) during six minutes walking test

SECONDARY OUTCOMES:
Thoracoabdominal mechanics | One week after the end of training
  The kinematic will be analyzed by optoelectronic plethysmograph during 30 seconds at rest, followed by 30 seconds after 3 minutes cycling without load, followed by 30 seconds after 30 minutes pedaling with load (25% of the calculated maximum watt).

OTHER OUTCOMES:
Anxiety and depression | One week after the end of training
  Measured by HADs Scale

CONTACTS AND LOCATIONS:
Overall Officials: Celso Carvalho, Dr., Study Director — Physiotherapy Departament of University of São Paulo
Locations (3):
- Brazil (3):
  - Physiotherapy Departament of University of São Paulo, São Paulo, São Paulo
  - FOFITO, São Paulo, São Paulo
  - Hospital das Clinicas, São Paulo, São Paulo